CLINICAL TRIAL: NCT06258785
Title: Effect of Pre-operative Tizanidine on Postoperative Urinary Retention After Sacrospinous Vaginal Vault Suspension: a Pilot Study
Brief Title: Effect of Tizanidine on Postoperative Urinary Retention After Sacrospinous Suspension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Claudia Paya Ten, Endeavor Health Urogynecology Fellow, Endeavor Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EH23-402
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Urinary Retention; Sacrospinous Vaginal Vault Suspension; Reconstructive Pelvic Surgery
MeSH Terms: interventions — tizanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tizanidine (Experimental): Tizanidine 2mg will be given preoperatively prior to scheduled sacrospinous ligament suspension
  Interventions: Drug: Tizanidine

INTERVENTIONS:
Drug: Tizanidine — Tizanidine 2mg will be given preoperatively prior to scheduled sacrospinous ligament suspension
  Other Names: Zanaflex

SUMMARY:
Postoperative urinary retention has been defined as the inability to void despite having fluid in the bladder during the postoperative period. Urinary retention after pelvic reconstructive surgery requiring indwelling catheter or self-catheterization usage occurs in approximately 30-60% of patients postoperatively. Our prior retrospective chart review reviewing postoperative urinary retention rates after pelvic reconstructive surgery demonstrated postoperative urinary retention after a sacrospinous vaginal vault suspension to be approximately 78.9%. Many women consider being discharged home with a Foley catheter to be a surgical complication and describe catheter use as the worst aspect of their surgery. Indwelling catheters are the leading cause of hospital-acquired urinary tract infections (UTIs), are often a source of embarrassment and inconvenience for patients, and often require additional office visits and healthcare utilization. Tizanidine is a muscle relaxant which can work to alleviate this spasm and, theoretically, prevent postoperative urinary retention. Tizanidine also works as an alpha-adrenergic receptor blocker which can increase smooth muscle relaxation around the urethra specifically and, theoretically, improve urine flow. Postoperative urinary retention is extremely common after pelvic reconstructive surgery involving a sacrospinous vaginal vault suspension and is extremely bothersome to patients. Tizanidine is a low-risk, well tolerated, cost-effective medication. No study to date has evaluated preoperative administration of tizanidine for postoperative urinary retention.

DETAILED DESCRIPTION:
Postoperative urinary retention has been defined as the inability to void despite having fluid in the bladder during the postoperative period. Urinary retention after pelvic reconstructive surgery requiring indwelling catheter or self-catheterization usage occurs in approximately 30-60% of patients postoperatively. Our prior retrospective chart review reviewing postoperative urinary retention rates after pelvic reconstructive surgery demonstrated postoperative urinary retention after a sacrospinous vaginal vault suspension to be approximately 78.9%.

Each patient after surgery undergoes a "voiding trial" where their voided volume is compared to their post-void residual volume. "Passing" a voiding trial has traditionally been defined as voiding a greater volume than the post-void residual volume. If the patient does not "pass" the voiding trial, the patient is characterized as having postoperative urinary retention and is discharged home with an indwelling catheter to prevent detrusor injury from bladder over-distention, pain and urinary tract infection.

Many women consider being discharged home with a Foley catheter to be a surgical complication and describe catheter use as the worst aspect of their surgery. Indwelling catheters are the leading cause of hospital-acquired urinary tract infections (UTIs), are often a source of embarrassment and inconvenience for patients, and often require additional office visits and healthcare utilization.

The leading hypotheses regarding the incidence of postoperative urinary retention after sacrospinous ligament suspension includes postoperative pain and pelvic floor muscle spasm leading to retention. The sacrospinous suspension includes a suture that is passed through the sacrospinous ligament and, therefore, through the coccygeus muscle with irritation of the pudendal nerve. The pelvic floor is a synergistic team of muscles that work together to support the pelvic organs and spasm of the coccygeus muscle, rather than an isolated muscle, can cause spasm of the entirety of the pelvic floor leading to retention. Tizanidine is a muscle relaxant which can work to alleviate this spasm and, theoretically, prevent postoperative urinary retention. Tizanidine also works as an alpha-adrenergic receptor blocker which can increase smooth muscle relaxation around the urethra specifically and, theoretically, improve urine flow.

Tizanidine is also frequently given for postoperative pain after sacrospinous ligament suspension and may act as an adjunct to a non-narcotic pain regimen to improve postoperative pain while reducing narcotic use after surgery. Postoperative buttock and posterior thigh pain are common symptoms after SSLF, with immediate pain reported in 6-84% of patients and persistent pain at 6 weeks occurring in 1-15%. Untreated acute postoperative pain has been shown to lead to increased morbidity and mortality. Pain is the most common reason for a postoperative unplanned hospital admission and poor postoperative pain control can lead to decreased ambulation, increased incidence of thromboembolism, and decreased inspiratory effort leading to postoperative pneumonia, therefore postoperative pain control is critical. In a country with rising narcotic-use and dependence, it is critical that we continue to explore non-narcotic alternatives for patients after surgery.

Postoperative urinary retention is extremely common after pelvic reconstructive surgery involving a sacrospinous vaginal vault suspension and is extremely bothersome to patients. Tizanidine is a low-risk, well tolerated, cost-effective medication. No study to date has evaluated preoperative administration of tizanidine for postoperative urinary retention.

ELIGIBILITY:
Inclusion Criteria:

* Sacrospinous ligament suspension (CPT 57282)

Exclusion Criteria:

* Age <18
* Planned combined cases with colorectal surgery, general surgery, or gynecology-oncology
* Known history of urinary retention
* Known contraindication to tizanidine

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This intervention is applicable for persons assigned female at birth undergoing sacrospinous ligament suspension for pelvic organ prolapse.
Enrollment: 20 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Paya Ten, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University Health System, Skokie, Illinois, United States

REFERENCES:
- [Background] Wang R, Won S, Haviland MJ, Von Bargen E, Hacker MR, Li J, Lefevre R. Voiding trial outcome following pelvic floor repair without incontinence procedures. Int Urogynecol J. 2016 Aug;27(8):1215-20. doi: 10.1007/s00192-016-2975-y. Epub 2016 Feb 17. PMID 26886553
- [Background] Geller EJ, Hankins KJ, Parnell BA, Robinson BL, Dunivan GC. Diagnostic accuracy of retrograde and spontaneous voiding trials for postoperative voiding dysfunction: a randomized controlled trial. Obstet Gynecol. 2011 Sep;118(3):637-642. doi: 10.1097/AOG.0b013e318229e8dd. PMID 21860294
- [Background] Willis-Gray MG, Wu JM, Field C, Pulliam S, Husk KE, Brueseke TJ, Geller EJ, Connolly A, Dieter AA. Is a Postvoid Residual Necessary? A Randomized Trial of Two Postoperative Voiding Protocols. Female Pelvic Med Reconstr Surg. 2021 Feb 1;27(2):e256-e260. doi: 10.1097/SPV.0000000000000743. PMID 31157716
- [Background] Pulvino JQ, Duecy EE, Buchsbaum GM, Flynn MK. Comparison of 2 techniques to predict voiding efficiency after inpatient urogynecologic surgery. J Urol. 2010 Oct;184(4):1408-12. doi: 10.1016/j.juro.2010.05.096. Epub 2010 Aug 19. PMID 20727543
- [Background] Pomajzl AJ, Siref LE. Postoperative Urinary Retention. 2023 Jul 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK549844/ PMID 31751034
- [Background] Elkadry EA, Kenton KS, FitzGerald MP, Shott S, Brubaker L. Patient-selected goals: a new perspective on surgical outcome. Am J Obstet Gynecol. 2003 Dec;189(6):1551-7; discussion 1557-8. doi: 10.1016/s0002-9378(03)00932-3. PMID 14710061
- [Background] Lovatsis D, Drutz HP. Safety and efficacy of sacrospinous vault suspension. Int Urogynecol J Pelvic Floor Dysfunct. 2002;13(5):308-13. doi: 10.1007/s001920200067. PMID 12355291
- [Background] Kondo W, Correa Leite GK, Fernandes R, Kamergorodsky G, Fin FR, Cordeiro Fernandes LF, Romeo A, Tessmann Zomer M. Useful Pelvic Retroperitoneal Neuroanatomy for Benign Gynecologic Surgery: A Cadaveric Dissection. J Minim Invasive Gynecol. 2021 Jan;28(1):20-21. doi: 10.1016/j.jmig.2020.05.013. Epub 2020 May 22. PMID 32450223
- [Background] Roshanravan SM, Wieslander CK, Schaffer JI, Corton MM. Neurovascular anatomy of the sacrospinous ligament region in female cadavers: Implications in sacrospinous ligament fixation. Am J Obstet Gynecol. 2007 Dec;197(6):660.e1-6. doi: 10.1016/j.ajog.2007.08.061. PMID 18060971
- [Background] Ghanavatian S, Derian A. Tizanidine. 2023 Aug 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK519505/ PMID 30137790
- [Background] Lovich-Sapola J, Smith CE, Brandt CP. Postoperative pain control. Surg Clin North Am. 2015 Apr;95(2):301-18. doi: 10.1016/j.suc.2014.10.002. Epub 2015 Jan 24. PMID 25814108
- [Background] Schug SA, Chong C. Pain management after ambulatory surgery. Curr Opin Anaesthesiol. 2009 Dec;22(6):738-43. doi: 10.1097/ACO.0b013e32833020f4. PMID 19606022
- [Background] Collins SA, Joshi G, Quiroz LH, Steinberg AC, Nihira MA. Pain management strategies for urogynecologic surgery: a review. Female Pelvic Med Reconstr Surg. 2014 Nov-Dec;20(6):310-5. doi: 10.1097/SPV.0000000000000134. PMID 25185632

RESULTS

PARTICIPANT FLOW:
Groups:
- Tizanidine: Patients will receive a single preoperative dose of tizanidine 2mg in the preoperative holding area on the day of scheduled sacrospinous ligament suspension.
Period: Overall Study
Arm/Group | Tizanidine
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tizanidine
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Smoking Status [Count of Participants; unit: Participants]
  Non-smoker | 14
  Prior smoker | 5
  Current smoker | 1
Menopausal Status [Count of Participants; unit: Participants]
  Pre-menopausal | 1
  Post-menopausal | 19
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28 (7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Urinary Retention
Description: Determine the postoperative urinary retention rates in patients undergoing a sacrospinous ligament suspension after postoperative administration of tizanidine. This will be determined immediately postoperative in the postoperative recovery room based on whether patients pass or fail their voiding trial described above. The result will be documented in electronic medical records and obtained from chart review.
Time Frame: Immediate postoperative evaluation (1 day)
Measure: Count of Participants; unit: Participants
Arm/Group | Tizanidine
Number analyzed (Participants) | 20
Participants | 11

2. Secondary Outcome: Average Postoperative Pain Score
Description: Determine average postoperative pain score after postoperative administration of tizanidine utilizing a 10-point Likert scale for pain (0 = no pain, 10 = extreme pain). This data will be obtained by electronic data pull and chart review.
Time Frame: Immediate postoperative evaluation (1 day)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tizanidine
Number analyzed (Participants) | 20
score on a scale | 3 (3)

3. Secondary Outcome: Number of Participants With Postoperative Unanticipated Healthcare Encounters
Description: Determine the number of participants with postoperative unanticipated healthcare encounters, including readmissions, office visits or emergency department visit within 30 days after surgery. This data will be collected via chart review.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tizanidine
Number analyzed (Participants) | 20
Participants | 1

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Tizanidine
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT06258785/Prot_SAP_000.pdf